CLINICAL TRIAL: NCT02635659
Title: The Effect of an Encapsulated Nutrient Mixture on Ileal Brake Activation: A Double-blind Randomized Study to Investigate the Effects on Body Weight, Food Intake and Satiety.
Brief Title: Proof of Concept Study; The Effect of an Encapsulated Nutrient Mixture on Ileal Brake Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: METC 143062
Record Dates: First submitted 2015-12-14; First posted 2015-12-21 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2015-12

CONDITIONS: Body Weight Decreased
Keywords: food intake, satiety, satiation, nutrients, ileal brake

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Encapsulated nutrients (Experimental): The investigational product will be a shot of sterile water (80 ml) mixed with a total of 21.6 grams encapsulate consisting of 13 grams of sucrose (60% of the total) encapsulated whey protein (<5% of total). On top of the encapsulated sucrose, 6.44 grams of casein (30% of total) encapsulated in whey protein (<5% of total) will be mixed with the shot of water. The micro-beats of encapsulated sucrose and casein are 150 µm and the ratio active (sucrose and casein) : whey is 95:5%, this means that the shot of water contains 13 grams of encapsulated sucrose, 6.44 grams of encapsulated casein and 1.3 grams of whey protein required for the encapsulation.
  Interventions: Other: Encapsulated nutrients
- Placebo (Placebo Comparator): The placebo has the same nutrient composition (e.g. 13 grams of sucrose and 6.44 grams of casein) as the active and will be equicaloric, and will also be mixed with a shot of sterile water (80 ml). The main difference of the placebo is that this nutrient mixture will be immediately released in the stomach, instead of being delivered to the ileum (active). This immediate release of the nutrient mixture is possible by using a different micro-encapsulation technique.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Encapsulated nutrients
  Arms: Encapsulated nutrients
Other: Placebo
  Arms: Placebo

SUMMARY:
Intraileal infusion of nutrients results in a reduction in food intake. A previous study by our group showed that both sucrose and casein infusion resulted in an increase in satiety and release of gastrointestinal peptides and a decrease in hunger and food intake. Encapsulating both nutrients, daily ingestion of this micro encapsulate and hereby releasing them in the distal small intestine could result in a chronic ileal brake activation. The obtained reduction in food intake and caloric intake could help overweight subjects to lose weight.

DETAILED DESCRIPTION:
Obesity and weight management Worldwide the incidence of overweight and obesity is rapidly increasing with negative impact on health and health care costs. The efficacy of the currently available treatments is relatively limited on the long term. So far, surgical intervention has been proven to be the only strategy to overcome severe obesity in the long-term. Furthermore, in a recent meta-analysis it was concluded that dietary supplements and exercise alone does not contribute to improved weight loss after caloric restriction diets. Therefore, it is important to develop new effective strategies that induce weight loss or help weight maintenance after weight loss. A promising mechanism for weight management is to activate the so called 'ileal brake'. Ileal brake The ileal brake refers to an intestinal feedback mechanism that is triggered by nutrients at a specific location in the small intestine, resulting not only in modulation of gastrointestinal secretions and motility but also of food intake and hunger. The ileal brake can be activated by ileal infusion of undigested lipid and recently it was found that ileal infusion of sucrose and casein suppresses food intake to the same extend as equicaloric amount of lipids8. In addition to the reduction of food intake, an increase in feelings of satiety and decrease in hunger was found. Since ileal brake activation seems to be a promising target for weight management strategies alternative nutrient delivery techniques have to be used. Several studies investigated the effects of nutrient infusion in all regions of the small intestine. However all studies used intestinal feeding catheters in order to infuse nutrients directly into the desired part of the small intestine. In order to investigate the effect of long-term ileal brake activation in overweight individuals, a different approach for nutrient delivery needs to be chosen. An alternative for distal small intestinal nutrient delivery via feeding catheters is encapsulation of nutrients. Encapsulation can be used to deliver nutrients to a specific intestinal location. By encapsulation, nutrients are covered/surrounded with an edible coating. This coating is defined as a thin layer of edible material applied to the surface of the nutrients. This provides a barrier against digestion in the stomach and the proximal parts of the small intestine. Comparable approaches have already been used for site-specific drug delivery. Two examples of systems able to deliver drugs to the ileo-colonic region are the ColoPulse system described by Schellekens et al. (2010) and the ileo-colonic delivery system described by Varum et al. (2013). Both methods are invented to accelerate drug release in the ileo-colonic region and use specific Eudragit® polymer coatings. Adjusting these polymer coatings results in a more proximal (ileum) delivery. However these techniques were developed for drug delivery. To activate the ileal brake it is preferred to use a completely food grade application. Another food grade approach to deliver nutrients to the distal small intestine is micro-encapsulation. This micro-encapsulation technique will be used in the present study to deliver a mixture of nutrients consisting mostly sucrose (60%) , casein (30%) in a shell of whey protein (10%) to the distal small intestine. The delivery method patented by AnaBio Technologies Ltd. (http://www.AnaBio.ie/) comprises an active component, encapsulated within a protein matrix of preferably whey protein. The mechanism by which their technique delivers the active to the preferred intestinal location is based on pH, surface porosity of the microspheres, and reaction to specific enzymes. These three parameters are used to design the micro-encapsulation beads to deliver the active ingredient to the preferred intestinal location (e.g. duodenum, jejunum or ileum). Furthermore the size of the micro-beads is important for intestinal transit time. AnaBio uses their data collected from human and animal studies to relate the size of the micro-beads to intestinal transit time, dose volume and physiological characteristics. The micro-bead size (micron range) can be chosen based on the population group and the required transit time, an average used size is 150 micron. The advantage of these small particles is that the particles can be mixed with a food product. The ratio active : encapsulated protein matrix is 95 : 5%. This means that if sucrose will be encapsulated 95% of the micro-bead is pure sucrose and 5% is whey protein. We know from our previous research8 that infusion with 13 grams of sucrose is able to activate the ileal brake. For the present study we will use a mixture of encapsulated sucrose microbeats (60%) and encapsulated casein microbeats (30%) in order to simulate the composition of a small mixed carbohydrate and protein rich meal. Efficacy small intestinal delivery AnaBio provided data (which cannot be shared due to IP applications) of four in vivo studies of which 3 were human studies and 1 pig study. In these studies the efficacy of their delivery method has been investigated. It can be concluded from these studies that the whey protein micro-encapsulation technique is a specific intestinal delivery method for specific to either the ileum (2 human studies and 1 pig study) or the jejunum (1 human study). Present study In the present study the effect of 6 weeks ileal brake activation on body weight, BMI and waist circumference will be investigated. It is hypothesized that 6 weeks ileal brake activation by delivery of an encapsulated nutrient mixture to the distal small intestine results in reduced body weight. This will be studied by daily ingestion of an encapsulated nutrient mixture (e.g. 60% sucrose and 30% casein encapsulated in 10% whey protein) either delivered to the distal small intestine (active) or stomach (placebo) before lunch and dinner for 6 weeks in a randomized, double blind parallel placebo controlled trial. This will be studied in the second phase of the study (phase 2). Pre intervention, study day 1 and 2 (SD1 and SD2), middle (SD4) and post (SD5) intervention period the efficacy of the to decrease food intake (>68 kcal) will be evaluated. It is unknown whether the ileal brake will be activated by the encapsulated nutrient mixture delivered to the distal small intestine (active) to the same magnitude as ileal brake activation by ileal sucrose and casein infusion. Therefore, we will study the ileal brake activation efficacy of the encapsulated nutrient mixture ingestion on ad libitum food intake. This will be done in the first phase of the study (phase 1). Pre-intervention the efficacy will be tested in a randomized placebo controlled cross over design. Within every subject the difference in ad libitum food intake after active or placebo ingestion will be studied. If the active encapsulated nutrient mixture does not result in a reduction of food intake the intervention will not start.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous examination, no gastrointestinal complaints can be defined.
* Age between 18 and 65 years. A higher age comes with a higher chance of comorbidities. These could influence our study outcomes and therefore this age range was chosen. This study will include healthy adult subjects (male and female). Women must be taking contraceptives (only needed in women with childbearing potential)
* BMI between 25 -30 kg/m2
* Normal Dutch eating habits eating three meals a day including breakfast as assessed by a validated questionnaire
* Voluntary participation
* Able to participate in the study, willing to give informed consent and to comply with the study procedures and restrictions

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided and documented by the principal investigator.
* Use of any medication, except oral contraceptives, which may interfere with this study (major interference with the execution of the experiment or potential influence on the study outcomes). This has to be decided and documented by the principle investigator.
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study, to be decided by the principle investigator, in the 90 days prior to the study.
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery) upon judgement of the principle investigator.
* Dieting (medically prescribed, diabetic and vegetarian)
* Pregnancy, lactation
* Excessive alcohol consumption (>20 alcoholic consumptions per week)
* Intention to stop smoking
* Self-admitted HIV-positive state
* Above average score (>2.26) on the restrained eating scale of the Dutch Eating Behaviour Questionnaire
* Reported unexplained weight loss or gain of >4 kg in the month prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Ileal brake activation and weight loss. | 43 days (measuring outcome at T=23 days and T=43 days)
  The difference in body weight before and after 6 weeks ileal brake activation by nutrient delivery to the distal small intestine (active; group 1) compared to nutrient mixture delivery to the stomach (placebo; group 2).

SECONDARY OUTCOMES:
Ileal brake and food intake. | 43 days (measuring outcome at T=23 days and T=43 days)
  To investigate whether intake of encapsulated nutrient mixture delivered in the distal small intestine (active) decreases the amount of food consumed during a subsequent ad libitum meal compared to encapsulated nutrient mixture delivered in the stomach (placebo) in time, analysed pre-, middle and post intervention.
Ileal brake and VAS scores. | 43 days (measuring outcome at T=23 days and T=43 days)
  To investigate whether intake of encapsulated nutrient mixture (active) increases satiation analysed by VAS-scores compared to placebo pre, middle and post intervention.

OTHER OUTCOMES:
Ileal brake and plasma GLP-1 level | 43 days (measuring outcome at T=23 days and T=43 days)
  To evaluate effects of 6 weeks encapsulated nutrient delivery to the distal small intestine (active) on GLP-1 plasma concentration compared to nutrient delivery to the stomach (placebo). This will be analysed by monitor blood glucose and insulin responses in time pre- and post-intervention.
Ileal brake and plasma glucose level | 43 days (measuring outcome at T=23 days and T=43 days)
  To evaluate effects of 6 weeks encapsulated nutrient delivery to the distal small intestine (active) on glucose plasma concentration compared to nutrient delivery to the stomach (placebo). This will be analysed by monitor blood glucose and insulin responses in time pre- and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: A.A.M. Masclee, MD, PhD, Principal Investigator — Maastricht University Medical Center (MUMC+)
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Anderson JW, Konz EC, Frederich RC, Wood CL. Long-term weight-loss maintenance: a meta-analysis of US studies. Am J Clin Nutr. 2001 Nov;74(5):579-84. doi: 10.1093/ajcn/74.5.579. PMID 11684524
- [Background] Batsis JA, Clark MM, Grothe K, Lopez-Jimenez F, Collazo-Clavell ML, Somers VK, Sarr MG. Self-efficacy after bariatric surgery for obesity. A population-based cohort study. Appetite. 2009 Jun;52(3):637-645. doi: 10.1016/j.appet.2009.02.017. Epub 2009 Mar 9. PMID 19501761
- [Background] Johansson K, Neovius M, Hemmingsson E. Effects of anti-obesity drugs, diet, and exercise on weight-loss maintenance after a very-low-calorie diet or low-calorie diet: a systematic review and meta-analysis of randomized controlled trials. Am J Clin Nutr. 2014 Jan;99(1):14-23. doi: 10.3945/ajcn.113.070052. Epub 2013 Oct 30. PMID 24172297
- [Background] Maljaars PW, Peters HP, Mela DJ, Masclee AA. Ileal brake: a sensible food target for appetite control. A review. Physiol Behav. 2008 Oct 20;95(3):271-81. doi: 10.1016/j.physbeh.2008.07.018. Epub 2008 Jul 21. PMID 18692080
- [Background] Maljaars PW, Peters HP, Kodde A, Geraedts M, Troost FJ, Haddeman E, Masclee AA. Length and site of the small intestine exposed to fat influences hunger and food intake. Br J Nutr. 2011 Nov;106(10):1609-15. doi: 10.1017/S0007114511002054. Epub 2011 Jun 7. PMID 21736790
- [Background] Maljaars J, Romeyn EA, Haddeman E, Peters HP, Masclee AA. Effect of fat saturation on satiety, hormone release, and food intake. Am J Clin Nutr. 2009 Apr;89(4):1019-24. doi: 10.3945/ajcn.2008.27335. Epub 2009 Feb 18. PMID 19225118
- [Background] van Avesaat M, Troost FJ, Ripken D, Hendriks HF, Masclee AA. Ileal brake activation: macronutrient-specific effects on eating behavior? Int J Obes (Lond). 2015 Feb;39(2):235-43. doi: 10.1038/ijo.2014.112. Epub 2014 Jun 24. PMID 24957485
- [Background] Shin HS, Ingram JR, McGill AT, Poppitt SD. Lipids, CHOs, proteins: can all macronutrients put a 'brake' on eating? Physiol Behav. 2013 Aug 15;120:114-23. doi: 10.1016/j.physbeh.2013.07.008. Epub 2013 Aug 1. PMID 23911804
- [Background] Schellekens RC, Stellaard F, Olsder GG, Woerdenbag HJ, Frijlink HW, Kosterink JG. Oral ileocolonic drug delivery by the colopulse-system: a bioavailability study in healthy volunteers. J Control Release. 2010 Sep 15;146(3):334-40. doi: 10.1016/j.jconrel.2010.05.028. Epub 2010 May 31. PMID 20621586
- [Background] Varum FJ, Hatton GB, Freire AC, Basit AW. A novel coating concept for ileo-colonic drug targeting: proof of concept in humans using scintigraphy. Eur J Pharm Biopharm. 2013 Aug;84(3):573-7. doi: 10.1016/j.ejpb.2013.01.002. Epub 2013 Jan 21. PMID 23348235
- [Background] Roza AM, Shizgal HM. The Harris Benedict equation reevaluated: resting energy requirements and the body cell mass. Am J Clin Nutr. 1984 Jul;40(1):168-82. doi: 10.1093/ajcn/40.1.168. PMID 6741850
- See also: WHO factsheet 311 — http://www.who.int/mediacentre/factsheets/fs311/en/